CLINICAL TRIAL: NCT05238116
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Safety and Efficacy of Nebulized PC945 When Added to Systemic Antifungal Therapy for the Treatment of Refractory Invasive Pulmonary Aspergillosis (OPERA-T Study)
Brief Title: Safety and Efficacy of PC945 (Opelconazole) in Combination With Other Antifungal Therapy for the Treatment of Refractory Invasive Pulmonary Aspergillosis (OPERA-T Study)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC_ASP_006; 2021-004554-32 (EudraCT Number); 2024-511281-36 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Refractory IPA
Keywords: Refractory IPA; invasive pulmonary aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PC945 (Experimental): PC945 dose, administered via nebulizer, twice daily
  Interventions: Drug: PC945
- Placebo (Placebo Comparator): PC945-placebo administered via nebulizer, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PC945 — Sterile aqueous liquid for Nebulization
  Arms: PC945
Drug: Placebo — Sterile aqueous liquid for Nebulization
  Arms: Placebo

SUMMARY:
To assess the safety and efficacy of nebulized PC945 in combination with systemic antifungal therapy for the treatment of refractory IPA

ELIGIBILITY:
Inclusion Criteria:

1. Participant has proven or probable IPA according to the modified 2019 European Organization for Research and Treatment of Cancer/ Mycoses Study Group Education and Research Consortium (EORTC/MSGERC) consensus definitions or according to the 2010 International Society for Heart and Lung Transplantation (ISHLT) consensus statements for the definitions of infections in cardiothoracic transplant recipients.
2. Participant's IPA has failed to respond to adequate antifungal therapy.

Exclusion Criteria:

1. Participant with a known or suspected concomitant medical condition or post-surgery complication that, in the opinion of the Investigator, may jeopardize adherence to the protocol requirements or impede the accurate measurement of efficacy or may be an unacceptable additional risk to the Participant should he/she participate in the study.
2. Participant who has previously received PC945.
3. Participant with a known history of allergy, hypersensitivity, or any previous serious reaction to any component of the PC945 or placebo formulations.
4. Participant who has recently received, is receiving or due to receive at any time during the study, an investigational medicinal agent that does not have any regulatory approved indications. Subjects who are participating in any other trials e.g., Observational, diagnostic or using medications with an approved indication may be allowed to participate after consultation with the sponsor on an individual basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Complete or Partial Overall Response | up to 12 weeks (Day 84)

SECONDARY OUTCOMES:
Time to Complete or Partial Overall Clinical Response | up to 12 weeks (Day 84)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (15):
  - Clinical Research Site, La Jolla, California
  - Clinical Research Site, Los Angeles, California
  - Clinical R Site, Los Angeles, California
  - Clinical Research Site, Sacramento, California
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Baltimore, Maryland
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, Minneapolis, Minnesota
  - Clinical Research Site, St Louis, Missouri
  - Clinical Research Site, The Bronx, New York
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Pittsburgh, Pennsylvania
  - Clinical Research Site 1, Houston, Texas
  - Clinical Research Site 2, Houston, Texas
  - Clinical Research Site, Madison, Wisconsin
- Argentina (5):
  - Clinical Research Site, Caba, Buenos Aires
  - Clinical Research Site, La Plata, Buenos Aires
  - Clinical Research Site, Caba, Buenos Aries
  - Clinical Research Site, Rosario, Santa Fe Province
  - Clinical Research Site, Mendoza
- Australia (2):
  - Clinical Research Site, Melbourne, Victoria
  - Clinical Research Site, Parkville, Victoria
- Austria (2):
  - Clinical Research Site, Graz, Styria
  - Clinical Research Site, Vienna
- Belgium (2):
  - Clinical Research Site, Brussels
  - Clinical Research Site, Leuven
- Brazil (6):
  - Clinical Research Site, Curitiba, Paraná
  - Clinical Research Site, Passo Fundo, Rio Grande do Sul
  - Clinical Research Site, Porto Alegre, Rio Grande do Sul
  - Clinical Research Site, Santa Maria, Rio Grande do Sul
  - Clinical Research Site, Jaú, São Paulo
  - Clinical Research Site, Santos, São Paulo
- Canada (2):
  - Clinical Research Site, Hamilton, Ontario
  - Clinical Research Site, Toronto, Ontario
- Clinical Research Site, Valparaíso, Chile
- Colombia (2):
  - Clinical Research Site, Montería, Departamento de Córdoba
  - Clinical Research Site, Cali, Valle del Cauca Department
- France (2):
  - Clinical Research Site, Paris
  - Clinical Research Site, Strasbourg
- Germany (2):
  - Clinical Research Site, Würzburg, Bavaria
  - Clinical Research Site, Frankfurt am Main, Hesse
- Greece (2):
  - Clinical Research Site, Athens
  - Clinical Research Site, Thessaloniki
- India (5):
  - Clinical Research Site, Bengaluru, Karnataka
  - Clinical Research Site 1, Pune, Maharashtra
  - Clinical Research Site 2, Pune, Maharashtra
  - Clinical Research Site, Hyderabad, Telangana
  - Clinical Research Site, New Delhi
- Israel (2):
  - Clinical Research Site, Haifa
  - Clinical Research Site, Ramat Gan
- Italy (5):
  - Clinical Research Site, Brescia, Lombardy
  - Clinical Research Site, Monza
  - Clinical Research Site, Naples
  - Clinical Research Site, Rome
  - Clinical Research Site, Siena
- South Korea (3):
  - Clinical Research Site, Daejeon
  - Clinical Research Site, Incheon
  - Clinical Research Site, Seoul
- Spain (5):
  - Clinical Research Site, Córdoba, Andalusia
  - Clinical Research Site, Barcelona, Catalonia
  - Clinical Research Site, Majadahonda, Madrid
  - Clinical Research Site, Granada
  - Clinical Research Site, Valencia
- Taiwan (3):
  - Clinical Research Site, Tapei City, Tapai
  - Clinical Research Site, Kaohsiung City
  - Clinical Research Site, New Taipei City
- Thailand (3):
  - Clinical Research Site, Khlong Luang, Changwat Pathum Thani
  - Clinical Research Site, Bangkok
  - Clinical Research Site, Khon Kaen
- United Kingdom (3):
  - Clinical Research Site, Harefield, Middlesex
  - Clinical Research Site, London
  - Clinical Research Site, Manchester

IPD SHARING:
Plan to Share IPD: No